CLINICAL TRIAL: NCT03075371
Title: Homeostatic and Non-homeostatic Processing of Food Cues in Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Heidelberg Medical Center (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Joe Simon, Principal Investigator, University of Heidelberg Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UHeidelbergMedCtr
Record Dates: First submitted 2017-02-28; First posted 2017-03-09 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Anorexia Nervosa; Healthy
MeSH Terms: conditions — Anorexia Nervosa | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intragastric glucose administration (Active Comparator)
  Interventions: Other: Glucose
- intragastric water administration (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Glucose — 75 g of glucose dissolved in 300 ml of water
  Arms: intragastric glucose administration
Other: Placebo — 300 ml of tap water
  Arms: intragastric water administration

SUMMARY:
The goal of the present study is to investigate metabolic gut-brain signaling and the neural correlates of distraction from visual food cues in patients with Anorexia nervosa and healthy controls.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is an eating disorder with high morbidity and lifetime mortality. This eating disorder is mainly characterized by restricted food intake despite a severely low body weight. Given the pronounced self-starvation in AN, the investigation of homeostatic food processing, and its interaction with the reward system is of great scientific interest. Previous research in AN patients has almost exclusively focused on cortical, non-homeostatic (e.g., reward related) food processing. Therefore, the primary aim of the present study is to investigate metabolic gut-brain signaling by focusing on the responsivity of the hypothalamus (i.e., the core region of homeostatic control) and the mesocorticolimbic reward system. A secondary aim is to study the interaction between the mesocorticolimbic reward system and the homeostatic (i.e., hypothalamus) system. Metabolic gut-brain signaling will be assessed by applying a single-blind, randomized, crossover design of intragastric infusion of glucose or water. This approach allows the study of gut-brain signaling to the hypothalamus and the reward system by controlling for sensory aspects of food intake (sight, smell, and taste) in AN patients and healthy controls. Furthermore, we will measure how cognitive strategies to control the desire for visual food cues (top-down control) affect the mesocorticolimbic and hypothalamic systems in AN patients differently than in healthy controls. The interaction between the hypothalamus and the mesocorticolimbic reward system will be investigated using an effective connectivity analysis. Functional magnetic resonance imaging with high spatial resolution and with an optimized protocol for the investigation of the hypothalamus and the mesocorticolimbic reward system will be used to study for the first time homeostatic and non-homeostatic food cue processing in AN patients.

ELIGIBILITY:
Inclusion Criteria:

* patients that meet the diagnostic criteria for AN (DSM-V criteria)
* Medically stable patients with a BMI < 17.5 kg/m² and > 13 kg/m²; Healthy controls with a BMI <25 kg/m² and >18.5 kg/m²
* Over Age of 18 years
* no other lifetimes or current medical illness that could potentially affect appetite or body weight
* right-handedness
* normal or corrected-to-normal vision

Exclusion Criteria:

* history of head injury or surgery
* history of neurological disorder
* severe psychiatric comorbidity (psychosis, bipolar disorder, substance abuse)
* smoking
* borderline personality disorder
* current psychotropic medication
* inability to undergo fMRI scanning (e.g. metallic implants, claustrophobia, Pacemakers)
* pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Resting state brain activity using fMRI | 35 min
  Functional brain imaging will be employed to assess metabolic gut-brain signaling during a single blind, randomized cross-over design of gastric glucose vs. water infusion.
Experimental fMRI task | 20 min
  Participants will be asked to either view food or nonfood images or to down-regulate their emotional response by distracting themselves from the stimuli by solving an arithmetic task.

SECONDARY OUTCOMES:
Analysis of hormonal satiety signaling | 30 min before scanning, 30 min after intragastric feeding, 60 min after intragastric feeding
  Blood is collected for the measurement of peripheral ghrelin. In total, three blood samples will be collected.
Self-report questionnaire regarding eating behavior (Dutch Eating Behavior Questionnaire) | 30 min
  Psychometric tests will be employed to assess eating behavior and eating disorder psychopathology (using the Dutch Eating Behavior Questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Joe Simon, Dr. Dipl. Psych., Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stopyra MA, Friederich HC, Lavandier N, Monning E, Bendszus M, Herzog W, Simon JJ. Homeostasis and food craving in obesity: a functional MRI study. Int J Obes (Lond). 2021 Nov;45(11):2464-2470. doi: 10.1038/s41366-021-00920-4. Epub 2021 Aug 17. PMID 34404907
- [Derived] Stopyra MA, Friederich HC, Monning E, Lavandier N, Bendszus M, Herzog W, Simon JJ. The influence of homeostatic mechanisms on neural regulation of food craving in anorexia nervosa. Psychol Med. 2021 Apr;51(6):1011-1019. doi: 10.1017/S0033291719003970. Epub 2020 Jan 14. PMID 31931900
- [Derived] Stopyra MA, Friederich HC, Sailer S, Pauen S, Bendszus M, Herzog W, Simon JJ. The effect of intestinal glucose load on neural regulation of food craving. Nutr Neurosci. 2021 Feb;24(2):109-118. doi: 10.1080/1028415X.2019.1600275. Epub 2019 Apr 15. PMID 30983543